CLINICAL TRIAL: NCT06521411
Title: A Pilot Study of a Subsidized and Culturally-adapted Community Supported Agriculture (CSA) Program
Brief Title: Pilot Subsidized and Culturally-adapted Community Supported Agriculture (CSA) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-00229-0
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Low-income Chinese American immigrant families with a focus on adults 18+ years in Brooklyn will participate in a culturally adapted systems -level program for improving diet.
  Interventions: Behavioral: CSA model

INTERVENTIONS:
Behavioral: CSA model — Community-supported agriculture (CSA) involves a community of individuals who support a farm and in return receive distributions of the farm's produce throughout the growing season. Culturally appropriate produce will be provided in subsidized weekly boxes for 20 weeks to community members at Brooklyn Grange Farm in Sunset Park at a fee of $5, which was determined to be acceptable by community members. Participants that receive SNAP benefits can use their EBT card to cover their $5. Education will be offered in the form of nutrition education, cooking tutorials, and farming information provided by staff at Brooklyn Grange.

SUMMARY:
This study aims to apply community-engaged methods to refine and implement a culturally adapted systems-level program for improving diet in low income, Chinese American immigrants. Guided by the regular partner engagement, The researchers have organically developed a systems-level program to bring a subsidized community-supported agriculture (CSA) model to the community in a way that is aligned with cultural values, and that includes culturally appropriate produce and nutrition education.

This is a single-site proof of concept pilot program that will be evaluated using a pre-post-design.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 years and over
* Currently living in Brooklyn
* Willing and able to provide consent

Exclusion Criteria:

• Unable to complete the baseline survey in English, Mandarin, or Cantonese

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Number of Different Vegetables Consumed | Baseline, Week 20
  Diet quality will be self-reported via a follow-up survey. The participant is presented with a list of 29 different vegetables - he/she is asked to select all of the vegetables in the list that was consumed in the past month.
Change in Diet Quality - Frequency | Baseline, Week 20
  Diet quality will be self-reported via a follow-up survey. Frequency (how often vegetables were consumed in the past month) is reported on a Likert scale: 1 = once a month, 2 = two or three times a month, 3 = once a week, 4 = more than once a week.
Change in Diet Quality - Quantity of Serving | Baseline, Week 20
  Diet quality will be self-reported via a follow-up survey. Quantity of Serving (how much is consumed at a time) is reported on a Likert Scale: 1 = less than ¼ cup, 2 = ¼ to ½ cup, and 3 = more than ½ cup.

SECONDARY OUTCOMES:
Change in Food Insecurity Score | Baseline, Week 20
  Food insecurity will be self-reported via a follow-up survey. The survey consists of 2 questions, reported on a Likert scale: 1 = often true, 2 = sometimes true, 3 = never true. The total range of score is 2-6; the higher the score, the lesser the insecurity.
Change in Social Cohesion Score | Baseline, Week 20
  Social cohesion will be self-reported via a follow-up survey. The survey consists of 3 questions, reported on a Likert scale: 0 = often, 1 = some of the time, 2 = hardly ever, 3 = never. The total score range is 0-9; the higher the score, the greater the sense of social cohesion.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Yi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Stella.Yi@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to stella.yi@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.